CLINICAL TRIAL: NCT01382355
Title: Prospective Donor Specific Antibody (DSA) Monitoring Protocol To Detect Patient Characteristics and /or Changes In Immunosuppression on the Development of De Novo Antibodies
Brief Title: Prospective Donor Specific Antibody (DSA) Monitoring Protocol
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Providence Health & Services (Other)
Collaborators: Washington State University (Other); Paul I Terasaki Foundation Laboratory (Unknown)
Responsible Party: Angela Maldonado PharmD, BCPS/Clinical Assistant Professor/Transplant Pharmacist, Providence Sacred Heart Medical Center
Other Study IDs: PDSAM 011
Record Dates: First submitted 2011-06-21; First posted 2011-06-27 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-08

CONDITIONS: Kidney Transplant; Kidney/Pancreas Transplant
Keywords: Kidney transplant; Kidney/Pancreas transplant; Antibody; Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1 ml aliquots of serum collected at specified time points
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Kidney transplant

SUMMARY:
Advances in transplant pharmacotherapy have led to improved one-year patient and graft survival in kidney transplant recipients, but have not translated to enhanced long-term survival. An explanation for the disparity in outcomes is the negative role of antibodies in transplant graft survival. There currently does not exist maintenance immunosuppression that targets antibodies and standard of practice aims at removing circulating donor specific antibodies upon detection of antibody mediated graft damage but not prior to the detection of rejection. There exists an insufficiency of data regarding patient and donor characteristics, changes in immunosuppression, the risk of viral donor and patient seropositivity and the risk of non-compliance on the development of antibodies. By measuring antibody levels in the blood at specific time periods after transplant, we may have a better understanding of what types of patients will develop antibodies, when these antibodies appear and how changes to transplant medications may affect antibodies.

The proposed project will examine the multifactorial risks associated with the development and appearance of donor-specific antibodies in the first year post-kidney transplant. The data collected will provide a historical perspective and preliminary pilot data to support a proposal for prospective antibody monitoring and to justify pre-emptively treating the antibodies in the absence of clinical signs of rejection.

DETAILED DESCRIPTION:
Organ transplantation is an effective treatment for several end-stage organ diseases. Preventing rejection of transplanted organs remains the premier challenge. According to the humoral theory, donor specific antibodies (DSA) are the major cause of chronic rejection and allograft loss. Despite this, and evidence that links human leukocyte antigen (HLA) antibodies to allograft dysfunction and loss, doubt remains about the cause-and-effect relationship and confirmation of this evidence is necessary to help facilitate change in transplant practice. Prospective monitoring for de novo DSA in the serum of patients who have received a transplant may allow for earlier detection, evaluation, and characterization of factors leading to the development of antibodies prior to the development of clinical manifestations of graft dysfunction.

The contribution of the major histocompatibility complex (MHC) Class I and Class II antibodies to transplant outcomes is well documented. However, there is emerging evidence that antibody mediated rejection and the severity of outcomes may involve proteins and antibodies that go beyond HLA Class I and II. A number of assays are available for testing for these additional antibodies and proteins but they are currently not used for widespread patient monitoring in part due to lack of data justifying their commercial use. This pilot study will prospectively evaluate for the presence and/or emergence of these unique antibodies, (I.E. MICA antigen, IgG3 and C1Q) in serial samples of serum, and confirm or reject the utility of incorporating these assays into routine patient monitoring which might provide earlier evidence of emerging rejection. Serum samples will be stored indefinitely for future kidney transplant research projects.

ELIGIBILITY:
Inclusion Criteria:

* Have received a living donor or deceased donor kidney/kidney pancreas transplant

Exclusion Criteria:

* Have not received a transplant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and females aged 18-70 years old receiving a living donor or deceased donor kidney or kidney/pancreas transplant
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who develop DSA within the first year post-transplant | 1 year
Risk factors for developing DSA | 1 year
  Patient demographics and immunosuppression regimen to be collected:
  Age at transplant Date of transplant Gender Race Cause of renal failure Donor type Repeat transplant (yes/no) Transplant current panel reactive antibody (PRA) Transplant flow crossmatch Previous crossmatch Serum creatinine at baseline DSA Class I/Class II, MICA, IgG3, C1Q Induction and maintenance immunosuppressant therapy Cytomegalovirus, BK virus, and Epstein Barr virus patient and donor seropositivity

SECONDARY OUTCOMES:
Change in allograft function at 1 year post-transplant compared to baseline (measured by Cockcroft-Gault) | 1 year
Incidence of patient survival at 1 year | 1 year
Proportion of patients who are DSA negative at 1 year | 1 year
Percent change of DSA from baseline to 1 year | 1 year
Proportion of Class I versus Class II detectable DSA that progress to antibody mediated rejection | 1 year
Incidence of allograft survival at 1 year | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Angela Q Maldonado, PharmD, Principal Investigator — Providence Sacred Heart Medical Center
Locations (1):
- Providence Sacred Heart Medical Center, Spokane, Washington, United States